CLINICAL TRIAL: NCT05784779
Title: Phase Ib/II Study to Evaluate the Efficacy and Safety of GH509 Versus Placebo in Patients With Nonalcoholic Steatohepatitis (NASH)/Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Phase Ib/II Study to Evaluate the Efficacy and Safety of GH509 Versus Placebo in Patients With NASH/NAFLD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 1Globe Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NASH-GH509-2
Record Dates: First submitted 2023-02-24; First posted 2023-03-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GH509 (Experimental)
  Interventions: Drug: GH509
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GH509 — Orally, once daily before bedtime (qhs)
  Arms: GH509
Drug: Placebo — Orally, once daily before bedtime (qhs)
  Arms: Placebo

SUMMARY:
This is a Phase Ib/II, randomized, double-blind, placebo-controlled, international multi-center clinical study to investigate the efficacy and safety of GH509 in subjects with NASH/NAFLD

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. ≥ 18 years of age and < 75 years old.
3. BMI ≥ 18 kg/m2.
4. Histologically confirmed NASH (defined as the presence of steatosis, inflammation, and ballooning) within 6 months prior to randomization with stage 2-3 fibrosis according to the NASH Clinical Research Network (CRN) classification OR NAFLD diagnosed by imaging assessment (MRI-PDFF ≥10% within 2 months prior to randomization).
5. ≤ 5% weight change within 6 months prior to randomization.
6. Diagnosed with T2DM.
7. For male or female patient of childbearing potential: Must agree to use contraception or take measures to avoid pregnancy during the study, and for 30 days (female) or 90 days (male) after the last dose of GH509/placebo.
8. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 5 days prior to randomization. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG.
9. Serum alanine transaminase (ALT) and serum aspartate transaminase (AST) ≤ 10×ULN within 14 days prior to randomization.
10. Serum creatinine <1.5×ULN within 14 days prior to randomization.
11. Platelets count ≥ 100,000/mm3 within 14 days prior to randomization.

Exclusion Criteria:

1. Subjects with a history of significant alcohol consumption for a period of more than 3 consecutive months any time within 1 year prior to screening.
2. Use of injected or oral antidiabetic agents within 3 months including: Thiazolidinediones; Subcutaneously administered agents; Sodium-glucose co-transporter 2 inhibitors
3. Patients with a history of hypoglycemia within 3 months before study enrollment.
4. Subject uses drugs historically associated with NASH/NAFLD for more than 2 weeks in the year prior to randomization.
5. Treatment with a non-stable dose of statins, fibrates, or proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor in 3 months prior to randomization.
6. LDL ≥190 mg/dL.
7. Treatment with a non-stable dose of drugs with potential anti-NASH/NAFLD effect in the 6 months prior to randomization.
8. Participated in a clinical research study with any investigational product being evaluated for the treatment of diabetes, weight loss, or NASH/NAFLD in the 6 months prior to randomization.
9. Subject is listed for orthotopic liver transplant (OLT) or has medical history of: biliary diversion, organ transplant/bone marrow transplant or undergoing immunosuppressive therapy, hepatocellular, pancreatic, thyroid carcinoma, multiple endocrine neoplasia syndrome type 2 (MEN 2) or other malignant disease.
10. Subject has prior or has planned bariatric surgery.
11. Subject had major surgery within 8 weeks prior to randomization, significant traumatic injury, or anticipation of need for major surgical procedure during the course of the study.
12. Presence of cirrhosis on liver biopsy.
13. Model for End-stage Liver Disease (MELD) score greater than 12.
14. Subject with clinical evidence of hepatic decompensation.
15. Subject has evidence of other forms of chronic liver disease:.
16. Acute cholecystitis or known biliary obstruction.
17. Acute or chronic pancreatitis or administration of total parenteral nutrition within 6 months prior to randomization.
18. Subject has gastrointestinal disorder(s) which would significantly impede the absorption of an oral agent.
19. Subject has concurrent severe infection including diagnoses of fever of unknown origin.
20. Clinically significant and uncontrolled cardiovascular disease within 12 months prior to randomization; cerebrovascular disease, grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication or grade II or greater peripheral vascular disease.
21. Subject with history of human immunodeficiency virus (HIV) infection.
22. Subject with known allergies to the study drug or any of its excipients.
23. Subject with an active, serious medical disease with likely life expectancy of less than 5 years.
24. Subject with active substance abuse, including alcohol and/or inhaled or injection drugs, in the year prior to randomization.
25. Subject has participated in an investigational new drug (IND) trial in the 30 days before randomization.
26. Subject has been previously exposed to GH509.
27. Unable or unwilling to swallow GH509/placebo daily.
28. Ineligibility for MRI.
29. Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
30. Subject has any other condition which would impede compliance or hinder completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Determine recommended Phase II dose (RP2D) | 12 weeks
  Determine the recommended Phase II dose (RP2D) of GH509, which is defined as the dose level that is well tolerated by patients
Change in liver fat content as assessed by MRI-PDFF | 12 weeks
  Proportion of patients achieving ≥30% hepatic fat reduction (assessed by MRI-PDFF) from baseline after 12 weeks of treatment

SECONDARY OUTCOMES:
Change in liver fat as assessed by MRI-PDFF | 12 weeks
  Change in percent of hepatic fat fraction assessed by MRI-PDFF from baseline after 12 weeks of treatment.
Proportion of MRI-PDFF responders | 12 weeks
  Proportion of patients achieving ≥30% hepatic fat reduction assessed by MRI-PDFF from baseline after 12 weeks of treatment
Change in liver enzymes as assessed by serum alanine aminotransferase (ALT) | 12 weeks
  Change in concentration of serum alanine aminotransferase (ALT) from baseline after 12 weeks of treatment.
Change in glycemic control as assessed by HbA1c | 12 weeks
  Change in percent of hemoglobin A1c (HbA1c) from baseline after 12 weeks of treatment.
Change in glycemic control as assessed by fasting blood glucose (FBG) | 12 weeks
  Change in concentration of fasting blood glucose (FBG) from baseline after 12 weeks of treatment.
Change in weight control as assessed by weight loss | 12 weeks
  Change in body weight from baseline after 12 weeks of treatment.
Tolerability and safety as assessed by incidence of adverse events | 16 weeks
  Number and percentage of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang, China